CLINICAL TRIAL: NCT04544241
Title: Cancer Survivorship and Caregiver Leadership Education for Clergy Wives and Widows
Brief Title: Cancer Leadership Training for Clergy Wives and Widows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1530494-1; 5U54MD007598-15 (NIH)
Record Dates: First submitted 2020-08-31; First posted 2020-09-10 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cancer; Patient Empowerment
Keywords: cancer; African American; church; clergy; leadership
MeSH Terms: conditions — Neoplasms; Patient Participation | interventions — Widowhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clergy Wives and Widows (Experimental): We will provide cancer survivorship and caregiving leadership education and activities for African American Clergy Wives and Widows by creating an educational partnership program aimed towards church-based health education on cancer survivorship and caregiving
  Interventions: Behavioral: Cancer Survivorship Leadership Training for Clergy Wives and Widows

INTERVENTIONS:
Behavioral: Cancer Survivorship Leadership Training for Clergy Wives and Widows — We will meet with Clergy Wives and Widows monthly for 2-3 hours over 10 months. These sessions will be delivered using innovative online format through Zoom over the ten months. During each meeting session, experienced community and academic leaders will present their expertise with relationship to cancer survivorship and caregiving. These individuals will have extensive experience in the particular area they are presenting in. In addition, allotted time will be given for discussion and group activities that can be performed virtually. To receive credit for completion of the training program, each participant must complete the training and deliver a group workshop. All clergy wives and widows will complete a demographic questionnaire, in addition to pre- and post- intervention questionnaires

SUMMARY:
Multiple cancer health disparities exist for underrepresented minority groups, such as higher late stage diagnoses and greater cancer-related deaths. Among African Americans, there is an increased cancer survivorship and caregiving burden, which necessitates more support and resources during these phases. The African American church has been evidenced to be a trusted source of resource and provide culturally competent care and contribute to decreasing these disparities. Importantly, the leadership of the African American churches are pivotal to the health and wellness of this population. One important leader is the clergy wife or widow, who is understudied but vital to the function of the church function and activities. The long-term goal of this proposed study is to develop a leadership training program for clergy wives and widows with emphasis on cancer survivorship and caregiving. The objective of this pilot project is to develop and test the Cancer Survivorship and Caregiver Leadership Education for Clergy Wives and Widows, with specific emphasis of cultural and spiritual considerations of African American cancer survivors and caregivers. The rationale for this project, is that African American clergy wives and widows can receive the necessary training to assist cancer survivors and caregivers in the management of physical, emotional, psychosocial, spiritual, and financial challenges. This study will be accomplished in four aims, which are 1) Develop skills and knowledge to perform an in-depth culturally sensitive need assessment and intervention map tailored for aging African American cancer survivors and caregivers, 2) To increase cancer survivorship and caregiving leadership education and activities for African American Clergy Wives and Widows, and 3) Enhance awareness of cancer-related health issues and its relationship to key determinants among aging cancer survivors and caregivers. This project is innovative in establishing a culturally and spiritually tailored intervention to develop the training of Clergy Wives and Widows to provide appropriate education for community dwelling African American survivors and caregivers. This research is significant because of its potential to inform cancer and caregiving related research and evidence-based practice for both health care professionals and community organizations and institutions to improve long term-health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Identify as either a clergy wife or widow
* Identify as African American and/or Black
* Live within the boundaries of Los Angeles County
* Be at least 18 years of age
* Speak and/or read English

Exclusion Criteria:

* Does not identify as a clergy wife or widow
* Does not self-identify as African American and/or Black
* Lives outside the boundaries of Los Angeles County
* Under the age of 18
* Unable to speak and/or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Cobb, PhD, Principal Investigator — Charles R. Drew University of Medicine & Science
Locations (1):
- Charles R. Drew University of Medicine & Science, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clergy Wives and Widows
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clergy Wives and Widows
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 22
Age, Continuous [Median (Full Range); unit: Years] | 59 [27 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 37
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Target Levels in Cancer Knowledge Using the Cancer Awareness Measurement Survey
Description: By comparison from baseline to post-intervention, there will be a 30% increase in the cancer awareness, risk factors, and screening among study participants.
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clergy Wives and Widows
Number analyzed (Participants) | 37
Participants | 20

2. Primary Outcome: Percentage of Participants Achieving Improvement in Mental Status and Wellness Using Depression, Anxiety, and Stress Survey
Description: By comparison from baseline to post-intervention, there will be a 30% increase in the awareness of depression, anxiety and stress among study participants.
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clergy Wives and Widows
Number analyzed (Participants) | 37
Participants | 25

3. Primary Outcome: Percentage of Participants Achieving Decreased Perceived Stigma Levels Using Cancer Stigma Scale
Description: By comparison from baseline to post-intervention, there will be a 30% decrease in cancer stigma among study participants.
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clergy Wives and Widows
Number analyzed (Participants) | 37
Participants | 30

4. Primary Outcome: Percentage of Participants Achieving Decreased Perceived Stress Using Caregiver Self-Assessment Questionnaire
Description: By comparison from baseline to post-intervention, there will be a 30% decrease in perceived stress regarding cancer caregiving among study participants.
Time Frame: 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clergy Wives and Widows
Number analyzed (Participants) | 37
Participants | 20

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Clergy Wives and Widows
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT04544241/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT04544241/ICF_001.pdf